CLINICAL TRIAL: NCT06035601
Title: An EHR-integrated Texting Platform to Promote Self-management in Women With Recurrent Urinary Tract Infections
Brief Title: EHR-integrated rUTI Texting Platform
Acronym: Urotrust
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Independence Blue Cross (Other)
Responsible Party: Principal Investigator, Lily Arya, Professor of OBGYN, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 853917
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: unnecessary antibiotics; self-management; digital platform; texting; implementation science; recurrent UTI; healthcare utilization; patient education
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistant extracting data on primary and secondary outcomes will be masked to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Electronic health record (EHR)-integrated texting platform (Experimental): Patients will be enrolled into a texting platform for the management of recurrent UTI.
  Interventions: Device: EHR-integrated texting platform (Urotrust)
- Usual care (Active Comparator): Patients will receive usual care through their providers.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: EHR-integrated texting platform (Urotrust) — * An evidence-based algorithm that provides symptom triage and clinical guidance during an episode of acute UTI
  * Evidence-based prevention education material on recurrent UTIs
  * 5 standing orders for urinalysis and urine culture in the EHR upon enrollment
  * Standard-of-care management for recurrent UTI
  Arms: Electronic health record (EHR)-integrated texting platform
Other: Usual care — • Standard-of-care management of recurrent UTI (phone calls and/or secure EHR messages for acute symptoms) and follow up visits as determined by patients and their providers.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to compare a texting platform to usual care for managing recurrent urinary tract infections (UTI).

The main question it aims to answer is:

• can a texting platform that integrates symptom triage and prevention education reduce the rate of unnecessary antibiotics for recurrent UTIs as compared to usual care?

Participants enrolled onto the texting platform will:

• receive evidence-based clinical guidance for the management of symptoms of UTI and receive educational videos on how to prevent UTIs. An important secondary outcome is to determine if the texting platform improves self-efficacy for the management of recurrent UTI.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Females who currently meet the criteria for recurrent UTIs
4. Age 18 years or older
5. Owns a mobile device with text messaging capability
6. Ability to read and write English
7. Currently receiving care from a provider in Penn Urogynecology or Penn Urology

Exclusion criteria:

1. History of known multidrug resistant UTIs
2. History of interstitial cystitis/bladder pain syndrome or current diagnosis of chronic pelvic pain
3. On continuous suppressive antibiotics currently
4. Currently pregnant or within 6 weeks of pregnancy
5. Transplant patient on immunosuppressive medication currently
6. Practice of chronic self-catheterization

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Rate of unnecessary antibiotics | 3 months
  Antibiotics prescribed for patients when 1) urine culture is negative and/or urine microscopy has pyuria < 10 WBC/HPF, 2) asymptomatic bacteriuria is present, or 3) there is no urine testing and no urinary symptoms.

SECONDARY OUTCOMES:
Patient self-efficacy | 3 months
  Stanford self-efficacy for managing chronic disease 6-item score (mean score range 1-10 with mean 1 indicating less self-efficacy)
Patient satisfaction: Patient Global Impression of Improvement score | 3 months
  Patient Global Impression of Improvement score (score range 1-7 with 1 indicating very much better)
Healthcare-related quality of life: EQ-5D-5L score | 3 months
  EQ-5D-5L score (score range 1-5 for each subscale with 1 indicating no problems)
Healthcare-related quality of life: Recurrent UTI Impact Questionnaire score | 3 months
  Recurrent UTI Impact Questionnaire score (score range 0-10 for each subscale with 0 indicating strongly disagree)
Healthcare utilization | 3 months
  Combined number of phone calls, secure messages, telehealth, and/or in-person visits per UTI episode
Antibiotic prescriptions | 3 months
  Number of antibiotic prescriptions given for UTI episodes
Patient medication compliance | 3 months
  Medication Adherence Self-Report Inventory score (score range 0-100 with 0 indicating no medication usage)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Agrawal S, Ikpeama N, Koelper N, Dokras A, Harvie H, Hamm RF, Dutcher L, Arya LA. A Randomized Trial of a Texting Platform for Recurrent Urinary Tract Infections. Urogynecology (Phila). 2026 Feb 2. doi: 10.1097/SPV.0000000000001770. Online ahead of print. PMID 41628883
- [Derived] Arya LA, Agrawal S, Ikpeama N, Harvie H, Feldman RH, Dutcher L. Implementing a Digital Platform for Recurrent Urinary Tract Infections. Urogynecology (Phila). 2025 Mar 1;31(3):183-193. doi: 10.1097/SPV.0000000000001604. Epub 2024 Nov 11. PMID 39527705